CLINICAL TRIAL: NCT03898830
Title: A Prospective, Controlled, Standardized, Multi-center, Single-treatment, Single-arm Evaluation of the Eon™ FR 1064 nm Device to Reduce Abdominal Fat With a 12-week Observation Interval to Assess Safe Fat Reduction
Brief Title: Eon™ FR Clinical Study Protocol 1064
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dominion Aesthetic Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0000000135
Record Dates: First submitted 2019-03-28; First posted 2019-04-02 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Fat Disorder
Keywords: Adipose tissue, abdominal
MeSH Terms: conditions — Lipid Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- eon™ FR 1064 nm device (Experimental): Patient will be treated with the eon™ FR 1064 nm device
  Interventions: Device: eon™ FR 1064 nm device

INTERVENTIONS:
Device: eon™ FR 1064 nm device — The subject treatment area - abdomen, was treated with the 1064 nm wavelength laser.

SUMMARY:
This study evaluates the treatment of subjects with the eon™ FR 1064 nm device in a single session to thermally induce apoptosis in adipose tissue.

DETAILED DESCRIPTION:
This study evaluates the treatment of subjects between 18-60 with the eon™ FR 1064 nm device in a single session to thermally induce apoptosis in adipose tissue in the abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 30 kg/m2 or less.
* Healthy male or female between the ages of 21 and 60.
* Had, at least 25 mm thickness adipose tissue on abdomen.
* Able to read, understand and sign the Informed Consent Form (ICF).
* Willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
* Willing to have limited sun exposure for the duration of the study, including the follow-up period.
* Willing to have photographs and ultrasound measurements taken of the treated area, which could be used de-identified in evaluations and could be used de-identified in presentations and/or publications.
* Female subjects were either post-menopausal, surgically sterilized, or used a medically acceptable form of birth control during the entire course of the study.
* Female subjects with child bearing potential were willing to take a urine pregnancy test and the result must be negative.
* Agreed to maintain their current diet and exercise habits and not be specifically trying to lose weight.

Exclusion Criteria:

* Aesthetic fat reduction procedure in the treatment area within the previous year.
* Age less than 21 or greater than 60 years old.
* Female subject pregnant or planning to become pregnant during the study duration,
* Had an infection, dermatitis or a rash in the treatment area.
* Had tattoos or jewelry in the treatment area.
* Had a history of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* Had a history of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* Had a history of a known bleeding disorder.
* Had a known photosensitivity to the study laser wavelength, history of ingesting. medications known to induce photosensitivity, or history of seizure disorders due to light.
* Had known collagen, vascular disease or scleroderma.
* Underwent a surgery or procedure in the treatment area within 6 months of treatment, which is still healing.
* Had underwent a fat reduction procedure in the treatment area within the past 12 months.
* Had a significant concurrent illness, such as insulin-dependent diabetes, peripheral vascular disease or peripheral neuropathy.
* Underwent systemic chemotherapy for the treatment of cancer.
* Used gold therapy for disorders such as rheumatologic disease or lupus.
* Participated in a study of another device or drug within three months prior to enrollment or during the study.
* As per the investigator's discretion, the subject had any physical or mental condition which might make it unsafe for the subject to participate in this study.
* Concurrent use of steroids or secondary rheumatoid drugs.
* Prior liposuction or a tummy tuck in the study area.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-12-08 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Photographic Evaluations as a Measure of Effectiveness | 12 weeks
  Photographs of the treatment area will be obtained at baseline and 12 weeks post treatment and be evaluated by blinded independent readers to correctly identify pre-treatment (baseline) photographs compared to 12 weeks post treatment photographs in order to determine effectiveness of device.

SECONDARY OUTCOMES:
Circumferential Measurements to Evaluate Reduction in Adipose Layer Thickness | 12 weeks
  Circumferential measurements of the treatment area will be completed and evaluated in comparison to the baseline results to determine the reduction in adipose layer thickness.
Ultrasound Measurement to Evaluate Reduction in Adipose Layer Thickness | 12 weeks
  Ultrasound of the treatment area will be performed and evaluated in comparison to the baseline results to determine the reduction in adipose layer thickness.
Subject Questionnaire to determine Subject Satisfaction | 12 weeks
  Subject Questionnaires will be completed by subjects at the end of study to determine the subject satisfaction with procedure.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Laser & Skin Surgery Center of Northern, Sacramento, California
  - Fiala Aesthetics, Altamonte Springs, Florida
  - Miami Dermatology & Laser Research, Miami, Florida

IPD SHARING:
Plan to Share IPD: No